CLINICAL TRIAL: NCT04954833
Title: Evaluating Visual Acuity and Initial Fit Performance of Two Soft Contact Lenses
Status: Completed | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6441
Record Dates: First submitted 2021-06-15; First posted 2021-07-08 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- TEST/CONTROL (Experimental): Eligible subjects will randomly be assigned to one of two unique sequences of the two lens types, Test/Control.
  Interventions: Device: EMO-200; Device: EMO-118
- CONTROL/TEST (Experimental): Eligible subjects will randomly be assigned to one of two unique sequences of the two lens types, Control/Test.
  Interventions: Device: EMO-200; Device: EMO-118

INTERVENTIONS:
Device: EMO-200 — TEST Lens
Device: EMO-118 — CONTROL Lens

SUMMARY:
This is a multi-center, randomized, controlled, double-masked, 2x2 cross-over, non-dispensing study to compare visual acuity and lens fit performance.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject's parents or legal guardians must read, understand, and sign the STATEMENT OF INFORMED CONSENT (Parental Permission Form and Authorization to Use and Disclose Medical Information). The subject must read (or be read to) and sign the CHILDREN'S ASSENT (Information and Assent Form) and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Between 7 and 12 (inclusive) years of age at the time of screening.
  4. Have normal eyes (i.e., no ocular medications or infections of any type).
  5. Have non-vertex corrected subjective spherical distance refraction in the range of -0.75 D to -4.50 D (inclusive) in each eye.
  6. Have refractive cylinder in the range of 0.00 D to -1.00 D (inclusive) in each eye with any degree of axis, by subjective sphero-cylindrical refraction.
  7. Have sphero-cylindrical best-corrected visual acuity of 0.04 logMAR (20/20-2) or better in each eye, and the difference of sphero-cylindrical best-corrected visual acuity between the two eyes is less than 0.20 logMAR (2 lines).
  8. Have < 1.50 D difference in subjective best-sphere refraction between the two eyes.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating.
  2. Have any systemic disease (e.g., Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g., rheumatoid arthritis), any underlying medical condition that makes subjects at risk of severe COVID complications, or other diseases, by parent of legal guardian's self-report, which are known to interfere with contact lens wear and/or participation in the study.
  3. Use of systemic medications (e.g., chronic steroid use) that are known to interfere with contact lens wear and/or participation in the study.
  4. Any current use of ocular medication (occasional use of re-wetting drops is allowed).
  5. Any previous or planned (during the course of the study) ocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
  6. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
  7. Current or recent (within 60 days from enrollment) wear of orthokeratology lenses.
  8. Current or recent (within 30 days from enrollment) rigid lens wearers.
  9. Immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  10. Children who are wards of the State or any other agency, institution, or entity.
  11. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, ocular hypertension, glaucoma, history of recurrent corneal erosions, aphakia, uveitis, severe keratoconjunctivitis sicca, keratoconus, keratoconus suspect, and pellucid marginal degeneration.
  12. Grade 3 or greater palpebral conjunctival observations or any other Grade 2 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, conjunctival injection) on the ISO 11980 classification scale.
  13. Any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear or subjects' participation in the study.
  14. Any central corneal scar.
  15. Any corneal distortion resulting from ocular diseases or previous hard or rigid gas permeable contact lens wear.
  16. Binocular vision abnormality, intermittent strabismus or strabismus.
  17. Pupil diameter under bright illumination is less than 2 mm in either eye.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- William J. Bogus, OD, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 60 subjects were enrolled in this study. Of those enrolled, 57 subjects were dispensed both study lenses and completed all study visits.
Groups:
- Test (EMO-200) \Control (EMO-118): Subjects randomized to this sequence received the Test lens during the first period and then received the Control lens during the second period
- Control (EMO-118) \Test (EMO-200): Subjects randomized to this sequence received the Control lens during the first period and then received the Test lens during the second period
Period: Period 1
Arm/Group | Test (EMO-200) \Control (EMO-118) | Control (EMO-118) \Test (EMO-200)
Started | 28 | 29
Completed | 28 | 29
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Test (EMO-200) \Control (EMO-118) | Control (EMO-118) \Test (EMO-200)
Started | 28 | 29
Completed | 28 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens
Groups:
- Total: All subjects dispensed a study lens
Arm/Group | Total
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.6 (1.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 24
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 2
  Black or African American | 1
  White | 54
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Monocular Distance Visual Acuity (logMAR)
Description: Visual acuity on logMAR (Logarithm of Minimal Angle of Resolution) scale was evaluated at distance (4 meters) under high luminance high contrast lighting condition using ETDRS (Early Treatment Diabetic Retinopathy Study) charts. Letter-by- letter results calculated the visual performance score for each chart read. LogMAR scores closer to zero, or below zero, indicate a better visual acuity. A logMAR visual performance score of 0.00 is equivalent to Snellen visual acuity of 20/20.
Time Frame: 10 minutes post lens insertion
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Groups:
- Test (EMO-200): Subjects that wore the Test lens in either the first or second period of the study.
- Control (EMO-118): Subjects that wore the Control lens in either the first or second period of the study.
Arm/Group | Test (EMO-200) | Control (EMO-118)
Number analyzed (Participants) | 57 | 57
Number analyzed (Eyes) | 114 | 114
logMAR | -0.00 (0.144) | -0.00 (0.140)
Statistical Analysis 1: Comparison: Test (EMO-200) vs Control (EMO-118); Test type: Non-Inferiority — A non-inferiority margin of 0.05 logMAR. A value of 0.05 logMAR is approximately 2.5 letters on the ETDRS chart; Mixed Model Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; LS Mean Difference = 0.01, 95% CI 2-sided [-0.01 to 0.02], Standard Error of Mean 0.006 — LS Mean difference was calculated as Test - Control

2. Secondary Outcome: Percentage of Subjects' Eyes With Acceptable Lens Fit
Description: Lens fit acceptance was assessed post lens fitting for each subject eye using a biomicroscope. Acceptable fit was a binary response where Y=1 if lens fit was deemed acceptable by the investigator and Y=0 otherwise. An unacceptable fit was observed if any of the following criteria were met: 1.) limbal exposure at primary gaze or with extreme eye movement, 2.) edge lift, 3.) excessive movement in primary and up gaze or 4.) insufficient movement in the three conditions- primary gaze, up gaze and Josephson push up. Time Frame 10 minutes post lens insertion
Time Frame: 10 minutes post lens insertion
Population: All subjects that were fitted at least one study lens
Measure: Number; unit: Percentage of acceptable lens fit
Units Other Than Participants: Eyes
Arm/Group | Test (EMO-200) | Control (EMO-118)
Number analyzed (Participants) | 57 | 57
Number analyzed (Eyes) | 114 | 114
Percentage of acceptable lens fit | 100 | 100
Statistical Analysis 1: Comparison: Test (EMO-200) vs Control (EMO-118); Test type: Non-Inferiority — A non-inferiority margin of 10% was used. A 10% of difference in the rate of lens fit acceptance is considered clinically significant; Bayesian hierarchical model; A 95% credible interval for the posterior mean difference between the Test and Control (Test - Control) was used to evaluate non-inferiority; Posterior mean difference of proportions = 0.000, 95% CI 2-sided [-0.009 to 0.010], Standard Deviation 0.0048 — Interval presented is a 95% Credible interval

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; The study duration for each subject is approximately 3 hours within 1 day.
Description: All subjects dispensed at least 1 study lens.
Arm/Group | Test (EMO-200) | Control (EMO-118)
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 0/57 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT04954833/Prot_SAP_000.pdf